CLINICAL TRIAL: NCT05491395
Title: Randomized Phase III Clinical Trial of Hypofractionated Radiotherapy in Breast Cancer Patients With Immediate Prosthetic Reconstruction: PROMART Trial
Brief Title: Hypofractionated Radiotherapy in Breast Cancer Patients With Prosthetic Reconstruction
Acronym: PROMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2022-06-13; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
Keywords: breast cancer, radiation therapy, hypofractionated, biomarkers
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Intervention Model Description: Arm Experimental: Post Mastectomy Hypofractionated Radiotherapy Arm No Intervention: Post Mastectomy Conventional Radiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post Mastectomy Hypofractionated Radiotherapy Arm (Experimental): Post Mastectomy Hypofractionated Radiotherapy Arm
  Interventions: Radiation: Hypofractionation
- Post Mastectomy Conventional Radiotherapy (No Intervention): Post Mastectomy Conventional Radiotherapy

INTERVENTIONS:
Radiation: Hypofractionation — Hypofractionation scheme will comprise 40 Gy in 15 fractions
  Arms: Post Mastectomy Hypofractionated Radiotherapy Arm

SUMMARY:
RATIONALE:

Radiotherapy (RT) can be indicated to patients submitted to breast-conserving surgery, but, despite the benefits, adjuvant RT can cause contracture generated by tissue fibrosis in patients with immediate prosthetic reconstruction, which could cause prosthesis loss. The biological explanation of this outcome is not fully understood, but recent advances in the analysis of patient-derived blood can contribute to establishing a connection of molecular alterations related to this clinical outcome.

There is not a consensus about using hypofractionated RT schemes for patients with BCS and breast reconstruction since no studies had investigated the reasons why some patients lose the prosthesis.

PURPOSE: This study will evaluate G3 toxicity rate in breast cancer patients with immediate prosthetic reconstruction, submitted to hypofractionated radiotherapy, analyzing capsular contracture, leakage, infection, and bad positioning in order to demonstrate the noninferiority of Hypo-RT with the conventional RT. Additionally, the molecular profile of blood samples will be investigated in order to find biomarkers related to inflammations processes and response to treatment.

DETAILED DESCRIPTION:
General aim: To evaluated if hypofractionated accelerated radiotherapy in patients with breast cancer undergoing immediate breast implant reconstruction surgery is non inferior to conventional radiotherapy.

Aim 1 (Primary objective): Assess the G3 toxicity rate - loss of the prosthesis (complication that requires surgical intervention: capsular contracture, leakage, infection, malpositioning).

Aim 2 (Specific secondary objectives):

* Compare local recurrence rate between two groups;
* Compare quality of life index between two groups using EORTC QLQ-C30 / EORTC QLQ-BR45 scales during treatment, after 6 and 12 months after treatment ending;
* Compare self-image differences between groups;
* Compare acute and late radiodermatitis rates by CTCAE 4.0;
* Analyse dosimetric planning differences considering the volumes of all breast and breast without prosthesis;
* Study inflammation molecular markers, which may indicate an increased risk of fibrosis;
* Evaluate the change in the profile of extracellular vesicles in patients treated with RT hypofractionated and conventional;
* Evaluate the change in EV collagen production after in vitro irradiation, using co-culture experiments with breast cells and fibroblasts.

ELIGIBILITY:
Inclusion Criteria:

* Women with confirmed histological diagnosis of invasive ductal carcinoma and lobular breast carcinoma;
* Radical mastectomy with immediate reconstruction with a prosthesis;
* Patients indicated for adjuvant RT;
* Any lymph node status;
* With or without adjuvant chemotherapy;
* ECOG performance status from 0-2;
* > 18 years old;
* Informed Consent Form applied before any study-specific procedure.

Exclusion Criteria:

* Another histological diagnosis than invasive ductal carcinoma or lobular carcinoma;
* Previous history of neoplasm and/or radiotherapy and/ or quimiotherapy before this study;
* Distant metastatic disease;
* Palliative treatment;
* Patients with scleroderma / systemic lupus erythematosus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Assess the G3 toxicity rate | 2 years
  loss of the prosthesis (complication that requires surgical intervention: capsular contracture, leakage, infection, malpositioning)

SECONDARY OUTCOMES:
Local recurrence | 5 years
  Compare local recurrence rate between two groups
Assessment of quality of life through the EORTC Questionnaires European Organization for Research and Treatment of Cancer, where a high or low score may suggest good quality of life depending on the domain of the questionnaire | 2 years
  Compare quality of life index between two groups using EORTC scales during treatment, after 6 and 12 months after treatment ending
Comparison of self-image using the EORTC Questionnaires European Organization for Research and Treatment of Cancer, where a high or low score may suggest good quality of life depending on the domain of the questionnaire | 5 years
  Compare self-image differences between groups
Compare acute and late radiodermatitis rates by Common Terminology Criteria for Adverse Events (CTCAE) 4.0 | 2 years
  Acute and late radiodermatitis rateswill be evaluated by CTCAE 4.0 scale, using the adverse event (AE) reporting. A grading (severity) scale is provided for each AE term.
Dosimetric analysis | 5 years
  Analyze dosimetric planning differences considering the volumes of all breast and breast without prosthesis
Inflammation markers screening - detection of cytokines with the CBA panel | 3 years
  Study inflammation molecular markers, which may indicate an increased risk of fibrosis. The cytokines present in the plasma will be evaluated using the Cytometric Beads Array technique with the CBA panel - Human Th1/Th2/Th17CBAKit which, through beads, is able to identify the expression of cytokines expressed by Th1, Th2 standard lymphocytes and Th17, including IL-2, IL-4, IL-6, IL-10, IL-17A, TNF e IFN-γ. After proper labeling, the immunophenotypic analyzes will be performed in a BD FAC Symphony flow cytometer.
Extracellular vesicles isolation and characterization | 4 years
  Evaluate the change in the profile of extracellular vesicles in patients treated with RT hypofractionated and conventional
Evaluate extracellular vesicles molecular profile | 4 years
  Evaluate the change in EV collagen production after in vitro irradiation, using co-culture experiments with breast cells and fibroblasts

CONTACTS AND LOCATIONS:
Overall Officials: Marcos D Mattos, MD, MS, Principal Investigator — Barretos Cancer Hospital; Gabriela B Salvador, BS, Study Chair — Barretos Cancer Hospital; Wanessa F Altei, PhD, Study Chair — Barretos Cancer Hospital; Lais L Almeida, MD, Study Chair — Barretos Cancer Hospital
Locations (1):
- Radiation Oncology Department, Barretos, São Paulo, Brazil

REFERENCES:
- [Background] Halsted WS. I. The Results of Operations for the Cure of Cancer of the Breast Performed at the Johns Hopkins Hospital from June, 1889, to January, 1894. Ann Surg. 1894 Nov;20(5):497-555. doi: 10.1097/00000658-189407000-00075. No abstract available. PMID 17860107
- [Background] Veronesi U, Saccozzi R, Del Vecchio M, Banfi A, Clemente C, De Lena M, Gallus G, Greco M, Luini A, Marubini E, Muscolino G, Rilke F, Salvadori B, Zecchini A, Zucali R. Comparing radical mastectomy with quadrantectomy, axillary dissection, and radiotherapy in patients with small cancers of the breast. N Engl J Med. 1981 Jul 2;305(1):6-11. doi: 10.1056/NEJM198107023050102. PMID 7015141
- [Background] Song SY, Chang JS, Fan KL, Kim MJ, Chang HP, Lew DH, Roh TS, Roh H, Kim YB, Lee DW. Hypofractionated Radiotherapy With Volumetric Modulated Arc Therapy Decreases Postoperative Complications in Prosthetic Breast Reconstructions: A Clinicopathologic Study. Front Oncol. 2020 Nov 17;10:577136. doi: 10.3389/fonc.2020.577136. eCollection 2020. PMID 33282731
- [Background] Liu L, Yang Y, Guo Q, Ren B, Peng Q, Zou L, Zhu Y, Tian Y. Comparing hypofractionated to conventional fractionated radiotherapy in postmastectomy breast cancer: a meta-analysis and systematic review. Radiat Oncol. 2020 Jan 17;15(1):17. doi: 10.1186/s13014-020-1463-1. PMID 31952507
- [Background] SBRT, Brazilian Society of Radiotherapy; Freitas NMA, Rosa AA, Marta GN, Hanna SA, Hanriot RM, Borges ABB, Gondim GRM, Pellizzon ACA, Veras IM, Almeida Junior WJ, Fernandez CRSHW, Batalha Filho ES, Castilho MS, Kuhnen FQ, Najas RMXF, Affonso Junior RJ, Leite ACC, Ribeiro HLM, Freitas Junior R, Oliveira HF. Recommendations for hypofractionated whole-breast irradiation. Rev Assoc Med Bras (1992). 2018 Sep;64(9):770-777. doi: 10.1590/1806-9282.64.09.770. PMID 30672995
- [Background] Van Poznak C, Somerfield MR, Bast RC, Cristofanilli M, Goetz MP, Gonzalez-Angulo AM, Hicks DG, Hill EG, Liu MC, Lucas W, Mayer IA, Mennel RG, Symmans WF, Hayes DF, Harris LN. Use of Biomarkers to Guide Decisions on Systemic Therapy for Women With Metastatic Breast Cancer: American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2015 Aug 20;33(24):2695-704. doi: 10.1200/JCO.2015.61.1459. Epub 2015 Jul 20. PMID 26195705
- [Background] Nimeus-Malmstrom E, Krogh M, Malmstrom P, Strand C, Fredriksson I, Karlsson P, Nordenskjold B, Stal O, Ostberg G, Peterson C, Ferno M. Gene expression profiling in primary breast cancer distinguishes patients developing local recurrence after breast-conservation surgery, with or without postoperative radiotherapy. Breast Cancer Res. 2008;10(2):R34. doi: 10.1186/bcr1997. Epub 2008 Apr 22. PMID 18430221
- [Background] Tramm T, Kyndi M, Myhre S, Nord S, Alsner J, Sorensen FB, Sorlie T, Overgaard J. Relationship between the prognostic and predictive value of the intrinsic subtypes and a validated gene profile predictive of loco-regional control and benefit from post-mastectomy radiotherapy in patients with high-risk breast cancer. Acta Oncol. 2014 Oct;53(10):1337-46. doi: 10.3109/0284186X.2014.925580. Epub 2014 Jun 24. PMID 24957550
- [Background] Kowal J, Arras G, Colombo M, Jouve M, Morath JP, Primdal-Bengtson B, Dingli F, Loew D, Tkach M, Thery C. Proteomic comparison defines novel markers to characterize heterogeneous populations of extracellular vesicle subtypes. Proc Natl Acad Sci U S A. 2016 Feb 23;113(8):E968-77. doi: 10.1073/pnas.1521230113. Epub 2016 Feb 8. PMID 26858453
- [Background] Yin Z, Yu M, Ma T, Zhang C, Huang S, Karimzadeh MR, Momtazi-Borojeni AA, Chen S. Mechanisms underlying low-clinical responses to PD-1/PD-L1 blocking antibodies in immunotherapy of cancer: a key role of exosomal PD-L1. J Immunother Cancer. 2021 Jan;9(1):e001698. doi: 10.1136/jitc-2020-001698. PMID 33472857
- [Background] Back M, Guerrieri M, Wratten C, Steigler A. Impact of radiation therapy on acute toxicity in breast conservation therapy for early breast cancer. Clin Oncol (R Coll Radiol). 2004 Feb;16(1):12-6. doi: 10.1016/j.clon.2003.08.005. PMID 14768750